CLINICAL TRIAL: NCT05295836
Title: Effects of Acute Glycerol Ingestion on Performance, Metabolic and Biochemical Markers in International Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Javier Martínez Noguera (Other)
Responsible Party: Sponsor-Investigator, Francisco Javier Martínez Noguera, Study coordinator (Investigator), Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CE102102
Record Dates: First submitted 2022-02-24; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Performance Enhancing Product Use; Change, Body Weight; Change, Body Temperature; Antioxidative Stress; Lactate Blood Increase; Thermal Sensation Disorders
Keywords: Power; Performance; Thermography; Metabolism; Endurance Sport; Ergogenic Aids; Oxygen uptake; Hydration; Hyperhydration
MeSH Terms: conditions — Body Weight Changes; Body Temperature Changes; Hyperlactatemia; Somatosensory Disorders; Water Intoxication | interventions — Glycerol

STUDY DESIGN:
Intervention Model Description: A randomized crossover study will be conducted, in which 4 international walkers will perform 3 different conditions: CON) water intake of 26 mL/kg/weight at 16°C; PLA) 26 mL/kg/weight + placebo at 28°C and GLY) intake of 1.2 g glycerol + 26 mL/kg/weight at 28°C.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): In this phase of the study, the rectangular test will be performed in conditions of 16°C and 25-30% humidity, intaking 26 mL/kg/body weight of water one and a half hours before the test.
- PLACEBO (PLA) (Placebo Comparator): In this intervention, subjects will perform the rectangular test at 28°C and 25-30% humidity, ingesting 26 mL/kg/body weight of water and placebo one and a half hours before the test.
  Interventions: Other: PLACEBO
- GLYCEROL (GLY) (Experimental): In this intervention, subjects will perform the rectangular test at 28°C and 25-30% humidity, ingesting 1.2 g + 26 mL/kg/body weight of water one and a half hours before the test.
  Interventions: Dietary Supplement: GLYCEROL

INTERVENTIONS:
Other: PLACEBO — Athletes will perform the rectangular test at a temperature of 28°C and ingested 26 mL/kg body weight + placebo one and half hours before the test.
  Arms: PLACEBO (PLA)
Dietary Supplement: GLYCEROL — Athletes will perform the rectangular test at a temperature of 28°C and ingested 26 mL/kg body weight + 1.2 g of glycerol one and half hours before the test.
  Arms: GLYCEROL (GLY)

SUMMARY:
This clinical study evaluates the acute effect of glycerol ingestion on performance (power output), weight, urine specific gravity, biochemical (antioxidants and lactate) and metabolic (indirect calorimetry) markers in international athletes in hot conditions. The investigators hypothesized that acute glycerol ingestion can prevent performance loss (power generated at submaximal intensity) in hot conditions. To justify this hypothesis, the investigators will measure the aforementioned markers, which could establish a cause-effect relationship between acute glycerol intake and decreased performance loss in hot conditions.

DETAILED DESCRIPTION:
All participants will be informed about the procedures and provide signed informed consent. The study will be conducted according to the guidelines of the Helsinki Declaration for Human Research and the protocol was approved by the Ethics Committee/Institutional Review Catholic University of Murcia (Code: CE091802).

Study design

This is a randomized crossover study. There are 3 types of intervention: water intake of 26 mL/kg/weight at 16°C (CON), 26 mL/kg/weight + placebo at 28°C (PLA) and intake of 1.2 g glycerol + 26 mL/kg/weight at 28°C (GLY). In addition, athletes will be instructed to take a individualized diet in relation to macronutrients (verified by dietary record) and they will follow their adjusted training schedule so that there would be no effect on the tests. Participants in both groups will be instructed not to consume supplements 3 weeks prior to the start of the study.

Procedures

Participants will visit the laboratory on five occasions. Visit 1 consists of a medical examination and a blood draw to determine health status. At visit 2, after a dinner the night before and a standard breakfast, an incremental test will be performed to determine the exercise zones in the rectangular test. At visits 3, 4 and 5, a record of the diet (individually set) will be performed regarding the former 7 days, followed by a rectangular treadmill test.

Visit 1:

Health status blood test: A general blood test will be performed. The blood will be drawn through a vein. (Fasting) Medical examination: A medical history of family and personal history, an electrocardiogram (ECG) at rest and a medical examination (auscultation, blood pressure, etc.) will be carried out to certify that the person is healthy and is not at risk to participate in the study. (Fasting)

Visits 2:

Incremental test with final ramp test will be performed on a cycle ergometer using a metabolic cart (Metalyzer 3B. Leipzig, Germany) to determine maximal fat oxidation zone (FatMax), ventilatory thresholds 1 (VT1) and 2 (VT2) and maximal oxygen consumption (VO2max). Participants will begin cycling at 35W for 2 min, increasing then by 35W every 2 min until RER>1.05, initializing then the final ramp (+35W·min-1) until exhaustion.

Visits 3:

The rectangular test will be performed on a treadmill using the speed values obtained in the incremental test (15 sets x 2 min at 95% with 2:30 recovery at 85% of maximum speed between sets). Cardiorespiratory variables (VO2, VCO2, VO2R, VE/VO2, VE/VCO2, VE/VCO2, respiratory coefficient, respiratory frequency, carbohydrate oxidation (CHO), fat oxidation (FAT), running economy and energy expenditure) will be determined in the 1st, 5th, 10th and 15th series.

For power measurement, each participant will wear the Stryd power meter, which is an inertial sensor (9.1 g) mounted on the foot, firmly attached to the shoe and according to the manufacturer's recommendations. The device stores at a sampling rate of 1 Hz the following variables: estimated power (PO), pace, cadence, leg sprint stiffness (LSS), form power, form power ratio, ground contact time (GCT), vertical oscillation, stride length. These variables will then be determined in the 1st, 5th, 10th and 15th series of the rectangular test. According to information from the Stryd team, the device is operational out of the box and should not require any calibration, accepting a measurement error of 3 percent. Participants will fill in their height and body mass prior to use, which is required for PO estimation. The firmware version that will be used is 2.1.16 (released in August 2020).

For lactate and antioxidant measurements, a Lactate Pro 2 meter and eBQC lab will be used on finger capillary blood at rest, after the 5th, 10th and after completion of the rectangular test.

For body temperature, the investigators will use an infrared thermographic camera (FLIR) to measure heat distribution (head, trunk, lower and upper limbs in both anterior and posterior aspects of the body).

Urine Samples Urine will be collected from the intake of water or water + glycerol or water + placebo until the start of the rectangular test and up to one hour after the rectangular test. The volume of urine excreted pre and post rectangular test will be recorded and the urine specific gravity will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Be an international athlete with the Spanish national athletics team.

Exclusion Criteria:

* Are smokers or regular alcohol drinkers,
* Have a metabolic, cardiorespiratory or digestive pathology or anomaly,
* Have an injury in the prior 6 months
* Are supplementing or medicating in the prior 2 weeks
* Have non-normal values in the blood analysis parameters.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Body weight | Throughout study completion, an average of 3 weeks
  Record body weight before and after the rectangular test
Urine specific gravity | Throughout study completion, an average of 3 weeks
  Record urine specific gravity by means a digital refractometer (Atago) before and after the rectangular test
Power output | Throughout study completion, an average of 3 weeks
  Record the power produced by means the stryd sensor (shoe) in the 1st, 5th, 10th and 15th series of the rectangular test
Body temperature | Throughout study completion, an average of 3 weeks
  Record body temperature by thermography of the head, trunk, and lower limbs, anterior and posterior in rest, after 5th and 10th series, and after completion of the rectangular test

SECONDARY OUTCOMES:
Lactate | Throughout study completion, an average of 3 weeks
  Record lactate in rest, after 5th and 10th series, and after completion of the rectangular test
Measurement of fast- and slow-acting antioxidants (Q1 and Q2) and total antioxidant capacity by a portable analyzer eBQC0101 | Throughout study completion, an average of 3 weeks
  Record the antioxidant markers in rest, after 5th and 10th series, and after completion of the rectangular test
Heart rate | Throughout study completion, an average of 3 weeks
  Record the heart rat in rest,1th, 5th, 10th and 15th series of the rectangular test
VO2 | Throughout study completion, an average of 3 weeks
  Record the oxygen uptake (L/min) in 1th, 5th, 10th and 15th series of the rectangular test
CO2 | Throughout study completion, an average of 3 weeks
  Record the carbon dioxide exhalation (L/min) in 1th, 5th, 10th and 15th series of the rectangular test
RER | Throughout study completion, an average of 3 weeks
  Record respiratory exchange ratio in 1th, 5th, 10th and 15th series of the rectangular test
VE | Throughout study completion, an average of 3 weeks
  Record ventilation (L/min) in 1th, 5th, 10th and 15th series of the rectangular test
FAT ox | Throughout study completion, an average of 3 weeks
  Record fat oxidation (g/h) in 1th, 5th, 10th and 15th series of the rectangular test
HC ox | Throughout study completion, an average of 3 weeks
  Record carbohydrate oxidation (g/h) in 1th, 5th, 10th and 15th series of the rectangular test
FR | Throughout study completion, an average of 3 weeks
  Record respiratory frequency (breaths/min) in 1th, 5th, 10th and 15th series of the rectangular test
EE | Throughout study completion, an average of 3 weeks
  Record energy expenditure (kcal/h) in 1th, 5th, 10th and 15th series of the rectangular test
V'E/V'O2 | Throughout study completion, an average of 3 weeks
  Record ventilatory equivalents for oxygen (L/min) in 1th, 5th, 10th and 15th series of the rectangular test
V'E/V'CO2 | Throughout study completion, an average of 3 weeks
  Record ventilatory equivalents for carbon dioxide (L/min) in 1th, 5th, 10th and 15th series of the rectangular test
VO2/R | Throughout study completion, an average of 3 weeks
  Record oxygen consumption relative to weight (mL/min/kg) in 1th, 5th, 10th and 15th series of the rectangular test
Cadence | Throughout study completion, an average of 3 weeks
  Record cadence (steps per minute) in 1th, 5th, 10th and 15th series of the rectangular test
Leg spring stiffness | Throughout study completion, an average of 3 weeks
  Record leg spring stiffness (kN/m) in 1th, 5th, 10th and 15th series of the rectangular test
Form power ratio | Throughout study completion, an average of 3 weeks
  Record form power ratio in 1th, 5th, 10th and 15th series of the rectangular test
Form power | Throughout study completion, an average of 3 weeks
  Record form power (W) in 1th, 5th, 10th and 15th series of the rectangular test
Ground contact time | Throughout study completion, an average of 3 weeks
  Record ground contact time (ms) in 1th, 5th, 10th and 15th series of the rectangular test
Vertical oscillation | Throughout study completion, an average of 3 weeks
  Record vertical oscillation (cm) in 1th, 5th, 10th and 15th series of the rectangular test
PO/R | Throughout study completion, an average of 3 weeks
  Record power output relative to weight (W/kg) in 1th, 5th, 10th and 15th series of the rectangular test

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Martínez Noguera, PhD, Study Chair — Research Center for High Performance Sport. Catholic University of Murcia
Locations (1):
- Research Center for High Performance Sport. Catholic University of Murcia, La Ñora, Murcia, Spain

REFERENCES:
- See also: Research Center for High Performance Sport. Catholic University of Murcia — http://investigacion.ucam.edu/vicerrectorado/ciard